CLINICAL TRIAL: NCT02595671
Title: B-slim, a Multi-source Digital Super Coach for Sustainable Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); iMinds (Industry); Brand New Health (Industry); Yorbody (Industry); Delhaize (Industry)
Responsible Party: Principal Investigator, Christophe Matthys, PhD, Prof. Christophe Matthys, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S57538
Record Dates: First submitted 2015-06-18; First posted 2015-11-03 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: Digital coaching; Sustainable weight loss; Self-determination theory; Obesity; Overweight; Diet; Physical activity
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Nutritionists

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Waiting Group (Active Comparator): Patients will not receive a treatment during the actual intervention. This group will receive the digital super coach as an incentive at the end of the trial.
  Interventions: Other: Waiting Group
- Conventional face to face PA & dietitian (Active Comparator): Participants will receive both dietary and physical activity advice. The advice is provided my medical trained staff (eg. dieticia, physiotherapist) according to a standardised protocol. The number of consultations are respectively three and four for diet and physcial activity.
  Interventions: Other: Conventional face to face PA & dietitian
- Digital Super Coach (Active Comparator): Only receive coaching via digital super coach.
  Interventions: Other: Digital Super Coach
- Digital Super Coach + minimal coaching (Active Comparator): Receive digital super coach and only have a few appointments with a physical activity coach and a dietitian.
  Interventions: Other: Digital Super Coach; Other: Digital Super Coach + minimal coaching

INTERVENTIONS:
Other: Digital Super Coach — Receive Digital Super Coach during 12 weeks
  Arms: Digital Super Coach; Digital Super Coach + minimal coaching
Other: Conventional face to face PA & dietitian — Receive 7 face-to-face contacts (dietary and physical activity advice)
  Arms: Conventional face to face PA & dietitian
Other: Digital Super Coach + minimal coaching — Receive 3 face-to-face contacts (dietary and physical activity advice)
  Arms: Digital Super Coach + minimal coaching
Other: Waiting Group — Receive Digital Super Coach during 12 weeks, after 12 weeks of no treatment
  Arms: Waiting Group

SUMMARY:
The purpose of this study is to carry out a field trial to evaluate the effectiveness and added value of the b-SLIM digital Super Coach in a convenient sample of overweight and obese adults.

DETAILED DESCRIPTION:
The purpose of this study is to carry out a field trial to evaluate the effectiveness of the b-SLIM digital Super Coach in a convenient sample of overweight and obese adults. The effectiveness will be evaluated at the individual level by means of a randomized trial. By combining or not combining the use of the b-SLIM digital Super Coach with a conventional physical activity and nutrition coaching, the effectiveness of the Super Coach of the (user-driven) 'Super Coach' compared to a conventional face to face weight loss program can be determined. Outcomes will be measured at the level of health behavior (i.e., physical activity and nutrition), body composition, physical fitness, psychosocial factors (e.g., motivation) and program adherence. The field trial will take place in Leuven (Belgium).

This study can be seen as a pilot trial. The central hypothesis of this field trial is that using the multi-source b-SLIM digital Super Coach will support and assist overweight and obese adults to change their health behavior (i.e., physical activity and nutrition) and to lose body weight by improving their self-control, self-determined motivation and attitude towards regular physical activity and healthy diet. The investigators will check if the Super Coach can be a valuable alternative for a conventional physical activity and nutrition coaching.

ELIGIBILITY:
Inclusion Criteria:

* Living in the region of Leuven
* Middle-aged (from 18 to 65 years)
* Having a body mass index between 29-34 kg/m²
* Having an e-mail address
* Having a personal computer

Exclusion Criteria:

* Suffering from a known physical (e.g., orthopedic limitations, stroke, etc.) and/or psychological (e.g., anorexia, bulimia, depression, etc.) disease or co-morbidity
* Intake of any medication with possible impact on body weight, endurance capacity
* Currently treated for diabetes (both Type 1 & 2).
* No sleepapneu has been determined during the last year.
* Having a history of systematic strength or endurance training (moderate to high intensity training more than once a week) in the year before the beginning of the trial
* Having a history of following a supervised dietary advice in the year before the beginning of the trial
* Having a history of bariatric surgery or any other malabsorption-related disease.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Weight Loss (Omron Weight Balance) | 12 weeks
  Weight loss measured pre & post intervenion

SECONDARY OUTCOMES:
Physical Activity - self evaluated | 12 weeks
  Physical activity measured by International Physical Activity Questionnaire
Physical Activity - objective measurement | 12 weeks
  Physical activity measured by ActiGraph
Food Litteracy | 12 weeks
  Food Litteracy measured by questionnaire
Dietary Pattern | 12 weeks
  Dietary pattern measured by the use of a Food Frequency Questionnaire
Body Composition - BIA | 12 weeks
  Using Bio-impediance Assessment to determine the fat and fatfree mass
Body Composition - 3D Scan | 12 weeks
  A 3D-scan will be used to evaluate phenotypic changes
Body Composition - Waist | 12 weeks
  Waist circumference measurement
Physical fitness | 12 weeks
  Use of the 6 minute walking test to evaluate the level of fitness of the participants
Motivation | 12 weeks
  Motivation to change lifestyle by use of a questionnaire
Social Support | 12 weeks
  social support will be measured by a questionnaire
Demographic factors | 12 weeks
  demographic factors will be measured by a questionnaire
Program adherence (24h food recall, compliance food pictures) | 12 weeks
  Adherence to the prescribed physical activity plan and dietary pattern
Shopping behavior | 12 weeks
  Shopping behavior (and potential changes) will be measured by use of the grocery fidelty card

OTHER OUTCOMES:
The usability experience | 3 months
  Usability and overall user experience of the Super Coach application

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Matthys, Prof. Dr., Study Chair — Department of Clinical and Experimental Medicine, KU Leuven; Jan Seghers, Prof. Dr., Study Chair — Physical Activity, Sports & Health (PASH) Research Group
Locations (1):
- University Hospital Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be discussed in the next steering committee

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Hurkmans E, Matthys C, Bogaerts A, Scheys L, Devloo K, Seghers J. Face-to-Face Versus Mobile Versus Blended Weight Loss Program: Randomized Clinical Trial. JMIR Mhealth Uhealth. 2018 Jan 11;6(1):e14. doi: 10.2196/mhealth.7713. PMID 29326093